CLINICAL TRIAL: NCT01638026
Title: Final Oocyte Maturation Via Administration of GnRH Agonists Followed By Luteal Support With hCG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Ronit Beck Fruchter, md, HaEmek Medical Center, Israel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: emc-0060-12-CTIL
Record Dates: First submitted 2012-07-08; First posted 2012-07-11 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Infertility
Keywords: Gnrh agonist
MeSH Terms: conditions — Infertility | interventions — Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gnrh agonist , hcg (Experimental): Gnrh agonist for final oocyte maturation, hcg for luteal support
  Interventions: Drug: TRIPTORELIN ACETATE, hCG

INTERVENTIONS:
Drug: TRIPTORELIN ACETATE, hCG — In the study group women will receive GnRH agonist (decapeptyl 0.2 mg) for oocyte maturation, followed by ovum pick-up which will be performed 35 hours later. Embryo transfer will be performed 48-72 hours after ovum pick-up. Luteal support will include HCG 1500 IU.

SUMMARY:
Study Objectives:

1. To prove that the use of GnHR agonist for final oocyte maturation results in a higher percentage of mature oocytes than the use of hCG.
2. To show an advantage in women's satisfaction in the proposed protocol versus the standard antagonist protocol In the study group women will receive GnRH agonist for oocyte maturation, followed by ovum pick-up which will be performed 35 hours later. Embryo transfer will be performed 48-72 hours after ovum pick-up. Luteal support will include HCG 1500 IU. Blood samples for BHCG, progesterone and estradiol will be obtained 14 days after embryo transfer.

DETAILED DESCRIPTION:
Final Oocyte Maturation via Administration of GnRH Agonists Followed By Luteal Support with hCG

The use of Gonadotropin-Releasing Hormone (GnRH) antagonists in in vitro fertilization (IVF) stimulation protocols holds many advantages over the long protocol with GnRH agonists. One of the advantages includes the ability to use GnRH agnosits for final oocyte maturation, thus minimizing the risk of ovarian hyperstimulation syndrome.

Study Objectives:

1. To prove that the use of GnHR agonist for final oocyte maturation results in a higher percentage of mature oocytes than the use of hCG.
2. To show an advantage in women's satisfaction in the proposed protocol versus the standard antagonist protocol

Inclusion criteria - patients who are eligible for in vitro fertilization using an antagonist protocol Exclusion criteria - patients diagnosed with hypogonadotrophic hypogonadism, sensitivity to any of the drugs used in the study A patient enrolled in the study who, as a result of ovarian stimulation, responds in a way that puts her in risk of developing ovarian hyperstimulation, will be ultimately excluded from the study. For the purpose of this study, this response includes estradiol levels higher than 2500 pg/ml, fifteen or more follicles over 12 mm in diameter, or any other case in which the treating physician has reason to suspect an eventual hyperstimulation reaction.

Study Protocol:

Informed consent will be obtained at the beginning of the treatment and up until the day of final oocyte maturation.

Oocyte stimulation in both groups will be achieved with recombinant FSH. Dose will be determined according to our department's protocol and response to previous treatments. GnRH antagonists will be added when leading follicle reaches 13-14 mm in diameter. Final oocyte maturation will be initiated when at least 2 follicles reach a diameter of 17 mm.

In the study group women will receive GnRH agonist (decapeptyl 0.2 mg) for oocyte maturation, followed by ovum pick-up which will be performed 35 hours later. Embryo transfer will be performed 48-72 hours after ovum pick-up. Luteal support will include HCG 1500 IU. Blood samples for BHCG, progesterone and estradiol will be obtained 14 days after embryo transfer. Prior to getting results from these tests, women will be asked to fill out a questionnaire regarding their satisfaction from the protocol protocol amendment: to add a prospective control group

We would like to add thromboelastography test. Our aim is to check whether triggering ovulation with GNRHa alters the clotting dynamics and reduce the risk for thromboembolic events.

Inclusion criteria:

IVF patients who are:

1. treated with the GNRH antagonist protocol
2. at low risk for OHSS
3. signed informed consent

Exclusion criteria:

IVF patients who:

1. are treated with the GNRH agonist protocol
2. infertile due to hypogonadotrophic hypogonadism
3. are at high risk of OHSS.

Study protocol:

Suitable patients would be offered to participate in the study and to sign informed consent. We will ask the participant to take 3 blood tests (5-8 ml blood each):

1. Before starting the hormonal treatment for ovulation induction.
2. During the hormonal treatment, 48-72 hours before ovum pickup.
3. At the day of the ovum pick up, about 36 hours after induction of final oocyte maturation using hCG or Gnrh agonist.

The study was approved by the local Ethics Committee. The thromboelastography test is available in the local hematologic laboratory. The cost of a single test is 50 NIS. We plan to recruit 50 patients.

Outcome:

Primary:

1. The change in the coagulation profile (the thromboelastogram) along the ovulation induction treatment.
2. The difference in the coagulation profile between the two different protocols, the GNRHa Vs the hCG.

Secondary:

The change in the coagulation profile in relation with:

1. estradiol levels
2. the number of oocytes
3. the number of embryos.
4. the achievement of pregnancy
5. the occurrence of OHSS.

ELIGIBILITY:
Inclusion Criteria:

* patients who are eligible for in vitro fertilization using an antagonist protocol

Exclusion Criteria:

* patients diagnosed with hypogonadotrophic hypogonadism, sensitivity to any of the drugs used in the study A patient enrolled in the study who, as a result of ovarian stimulation, responds in a way that puts her in risk of developing ovarian hyperstimulation, will be ultimately excluded from the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2012-09; Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
fertilization rate | 4 weeks

SECONDARY OUTCOMES:
satisfaction, no. of oocyte, pregnancy rate, no. of embryos, quality of embryos | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hemek medical centre, Afula, Israel